CLINICAL TRIAL: NCT04234568
Title: A Phase I Trial of Triapine and Lutetium Lu 177 Dotatate in Combination for Well-Differentiated Somatostatin Receptor-Positive Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs)
Brief Title: Testing the Addition of an Anti-cancer Drug, Triapine, to the Usual Radiation-Based Treatment (Lutetium Lu 177 Dotatate) for Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-00170; NCI-2020-00170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-CIRB-10388-PMC; 10388 (Other: Ohio State University Comprehensive Cancer Center LAO); 10388 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2020-01-17; First posted 2020-01-21 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Digestive System Neuroendocrine Neoplasm; Metastatic Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Specimen Handling; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lutetium Lu 177 dotatate, triapine) (Experimental): Patients receive lutetium Lu 177 dotatate IV for 30 to 40 minutes on day 1 of each cycle and triapine PO on days 1 throughout 14 of each cycle. Cycles repeat every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan or MRI scan throughout the trial. Patients undergo blood specimen collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lutetium Lu 177 Dotatate; Procedure: Magnetic Resonance Imaging; Drug: Triapine

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium (177Lu) Oxodotreotide; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Triapine — Given PO
  Other Names: 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; 3-AP; 3-Apct; OCX-0191; OCX-191; OCX191; PAN-811

SUMMARY:
This phase I trial studies the side effects and best dose of triapine when given together with lutetium Lu 177 dotatate in treating patients with neuroendocrine tumors. Triapine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radioactive drugs, such as lutetium Lu 177 dotatate, may carry radiation directly to tumor cells and not harm normal cells. Giving triapine and lutetium Lu 177 dotatate together may work better to treat patients with neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and to determine the recommended phase 2 dose (RP2D) of lutetium Lu 177 dotatate in combination with triapine.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at 2, 4, 6, and 8 months post therapy in dose escalation cohort.

III. To determine the best overall response rate (ORR) by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 in dose expansion cohort.

IV. To measure duration of response (DOR) associated with the combination. V. To evaluate progression-free survival (PFS), 24-month PFS, and overall survival (OS).

CORRELATIVE OBJECTIVES:

I. Measure baseline 68 gallium-dotatate (or copper 64 dotatate) biodistribution.

II. Evaluate oral triapine plasma pharmacokinetics and corresponding methemoglobin level by venous blood gas proportion.

III. Collect blood at baseline and at disease progression to correlate result with clinical outcome. (NOTE: originally this blood was collected to analyze hPG80 but will now the frozen blood samples will be biobanked for future correlative analysis) IV. Describe the tumor molecular profile using whole exome sequencing (WES), as well as ribonucleic acid sequencing (RNAseq) by the National Clinical Laboratory Network (NCLN), and correlate it with treatment outcome.

V. Collect plasma for circulating deoxyribonucleic acid (DNA) (ctDNA) assessment.

VI. Assess the effect of triapine on single deoxyribonucleoside concentrations by a liquid chromatography-mass spectrometry (LC/MSMS) assay in baseline (pre-treatment) and disease progression blood samples (processed to plasma).

OUTLINE: This is a dose-escalation study of triapine followed by a dose-expansion study.

Patients receive lutetium Lu 177 dotatate intravenously (IV) for 30 to 40 minutes on day 1 of each cycle and triapine orally (PO) on days 1 throughout 14 of each cycle. Cycles repeat every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) scan throughout the trial. Patients undergo blood specimen collection on study.

Patients are followed up every 3 months for 24 months from the time of enrollment. Patients removed from study for unacceptable adverse event(s) are followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, histologically confirmed well-differentiated neuroendocrine tumor with positive dotatate scan (gallium-68 or copper-64) within 6 months. Lesions on dotatate scan (gallium-68 or copper-64 dotatate scan) will be considered positive if the maximum standard uptake value (SUVmax) is > 2 times SUV mean of normal liver parenchyma
* Failure of at least one prior systemic cancer treatment, including somatostatin analogs
* Patients must have progressive disease based on RECIST criteria, version 1.1 evidenced with CT scans/MRI obtained within 24 months from enrollment
* Patients must have measurable disease per RECIST 1.1
* No prior exposure to peptide receptor radionuclide therapy
* Recovered from adverse events of previously administered therapeutic agents to grade 1 or less toxicity according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
* Archival tissue no longer than 6 months old should be present, otherwise baseline research biopsy is needed for WES
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of triapine in combination with lutetium Lu 177 dotatate in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1, or 2 (Karnofsky >= 60%)
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 3 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Glomerular filtration rate (GFR) >= 50 mL/min using Cockcroft-Gault method
* Hemoglobin >= 8.0 g/dL
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen, in the opinion of the enrolling physician, are eligible for this trial
* Pregnancy precaution: Men and women should avoid pregnancy for seven months after the date of their last treatment with lutetium Lu 177 dotatate. It is noteworthy that beta-human chorionic gonadotropin (HCG) may be secreted by a small percentage of neuroendocrine tumors (NETs), such that, in addition to being a pregnancy marker, it also is a tumor marker. Consequently, NET female patients with positive beta-HCG (> 5 mIU/mL) at baseline can be eligible to enter the study and receive treatment if pregnancy can be excluded by lack of expected doubling of beta-HCG and negative pelvic ultrasound. Normally, in pregnant subjects beta-HCG doubles every 2 days during the first 4 weeks of pregnancy and every 3.5 days by weeks 6 to 7. Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral ovariectomy) or is not postmenopausal (defined as amenorrhea > 12 consecutive months, and for women on hormone replacement therapy, only with a documented plasma follicle-stimulating hormone [FSH)] level > 35 mIU/mL). Even women who are using oral, implanted, or injected contraceptive hormones, an intrauterine device (IUD), or barrier methods (diaphragm, condoms, spermicidal) to prevent pregnancy, are practicing abstinence or where the partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential. Postmenopausal women who have fertilized eggs implanted are also considered to be of childbearing potential. Acceptable methods of contraception may include total abstinence at the discretion of the Investigator in cases where the age, career, lifestyle, or sexual orientation of the patient ensures compliance. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Reliable contraception (hormonal or barrier method of birth control; abstinence) should be maintained throughout the study and for 7 months after study treatment discontinuation. All women of childbearing potential and male partners must use a double-barrier method of birth control or practice continuous abstinence from heterosexual contact throughout the study and for seven months after the end of the last treatment
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have had major surgical procedures in the prior 6 weeks
* Patients with an inability to swallow oral medications or gastrointestinal disease limiting absorption of oral agents
* Patients who have received prior external beam radiotherapy to more than 50% of bone marrow, as determined by a radiation medicine physicist who will calculate the volume of bone marrow exposure in prior radiotherapy portals divided by the volume of total bone marrow harboring tissues. This ratio must be less than 50 percent
* Uncontrolled congestive heart failure (New York Heart Association [NYHA] III, IV)
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to triapine or lutetium Lu 177 dotatate
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection; symptomatic decompensated congestive heart failure; unstable angina pectoris; cardiac arrhythmia; and known inadequately controlled hypertension
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because triapine is a ribonucleotide reductase (RNR) inhibitor and lutetium Lu 177 dotatate is a peptide receptor radionuclide therapy with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with triapine and lutetium Lu 177 dotatate, breastfeeding should be discontinued if the mother is treated with triapine and lutetium Lu 177 dotatate and for 2.5 months following the last treatment
* Discontinue long-acting somatostatin analogs (e.g., long-acting octreotide) for at least 4 weeks prior to initiating lutetium Lu 177 dotatate. Long-acting somatostatin analog will be allowed to continue if patient has history of carcinoid syndrome and requires long-acting somatostatin analog for control of his/her functional syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2026-03-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Arnold, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (11):
- United States (11):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were consented and enrolled to the study but were subsequently discovered to be screen failures. They did not receive study treatment or get assigned to an arm.
Groups:
- Escalation Phase Dose Level 1 (100mg Triapine); Escalation Phase Dose Level 2 (150mg Triapine); Escalation Phase Dose Level 3 (200mg Triapine); Expansion Phase Dose Level 1 (100mg Triapine); Expansion Phase Dose Level 2 (150mg Triapine): Patients receive lutetium Lu 177 dotatate IV for 30 to 40 minutes on day 1 of each cycle and triapine PO on days 1 throughout 14 of each cycle. Cycles repeat every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan or MRI scan throughout the trial. Patients undergo blood specimen collection on study.
  Biospecimen Collection: Correlative studies
  Computed Tomography: Undergo CT
  Lutetium Lu 177 Dotatate: Given IV
  Magnetic Resonance Imaging: Undergo MRI
  Triapine: Given PO
Period: Overall Study
Arm/Group | Escalation Phase Dose Level 1 (100mg Triapine) | Escalation Phase Dose Level 2 (150mg Triapine) | Escalation Phase Dose Level 3 (200mg Triapine) | Expansion Phase Dose Level 1 (100mg Triapine) | Expansion Phase Dose Level 2 (150mg Triapine)
Started | 3 | 11 | 1 | 2 | 14
Completed | 3 | 11 | 1 | 2 | 14
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escalation Phase Dose Level 1 (100mg Triapine) | Escalation Phase Dose Level 2 (150mg Triapine) | Escalation Phase Dose Level 3 (200mg Triapine) | Expansion Phase Dose Level 1 (100mg Triapine) | Expansion Phase Dose Level 2 (150mg Triapine) | Total
Number analyzed (Participants) | 3 | 11 | 1 | 2 | 14 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 10 | 0 | 1 | 11 | 24
  >=65 years | 1 | 1 | 1 | 1 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 1 | 9 | 13
  Male | 2 | 9 | 1 | 1 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 11 | 1 | 2 | 12 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 2
  White | 3 | 10 | 1 | 2 | 12 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 11 | 1 | 2 | 14 | 31
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status measures effect of symptoms and is based on a scale with grades from 0 to 5, with 5 representing the worst outcome. Below are descriptions for the two grades represented in the study's baseline population.
  Grade 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    Grade 0 | 2 | 9 | 0 | 0 | 10 | 21
    Grade 1 | 1 | 2 | 1 | 2 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Triapine and Recommended Phase 2 Dose (RP2D)
Description: The MTD and RP2D will be estimated using isotonic regression based on observed dose limiting toxicity from all patients enrolled in the phase 1 portion and expansion cohort. All patients who received study drugs will be included in the safety analysis.
Time Frame: 8 weeks (56 days)
Population: One patient in the expansion phase was not evaluable for dose limiting toxicity or for MTD determination
Measure: Number; unit: milligrams
Groups:
- Escalation Phase; Expansion Phase: Patients receive lutetium Lu 177 dotatate IV for 30 to 40 minutes on day 1 of each cycle and triapine PO on days 1 throughout 14 of each cycle. Cycles repeat every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan or MRI scan throughout the trial. Patients undergo blood specimen collection on study.
  Biospecimen Collection: Correlative studies
  Computed Tomography: Undergo CT
  Lutetium Lu 177 Dotatate: Given IV
  Magnetic Resonance Imaging: Undergo MRI
  Triapine: Given PO
Arm/Group | Escalation Phase | Expansion Phase
Number analyzed (Participants) | 15 | 15
milligrams | 150 | 150

2. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: DLTs will be summarized descriptively at each dose level. Will be summarized based on Common Terminology Criteria for Adverse Events version 5.0. The maximum grade of toxicity for each adverse event category of interest will be recorded for each patient and the summary results will be tabulated by category and grade. Will describe all serious (>= grade 3) toxicity events on a patient-by-patient basis. Frequency and incidence tables of toxicity and adverse events will be generated in the overall patient group and by dose level depending on patient enrollment.
Time Frame: 8 weeks (56 days)
Population: One patient from the expansion phase was not evaluable for DLTs.
Measure: Number; unit: participants
Arm/Group | Escalation Phase Dose Level 1 (100mg Triapine) | Escalation Phase Dose Level 2 (150mg Triapine) | Escalation Phase Dose Level 3 (200mg Triapine) | Expansion Phase Dose Level 1 (100mg Triapine) | Expansion Phase Dose Level 2 (150mg Triapine)
Number analyzed (Participants) | 3 | 11 | 1 | 2 | 13
participants
  Grade 4 Neutropenia | 0 | 2 | 0 | 0 | 5
  Grade 5 Cardiac Arrest | 0 | 0 | 1 | 0 | 0
  Grade 3 Anemia | 0 | 0 | 0 | 1 | 0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR will be estimated along with 95% exact binomial confidence interval.
Time Frame: From the start of the treatment until disease progression/recurrence, assessed up to 24 months
Population: One patient from the escalation phase dose level 3, and two patients from the expansion phase dose level 2 were unevaluable for overall response.
Measure: Number; unit: percentage of participants
Arm/Group | Escalation Phase Dose Level 1 (100mg Triapine) | Escalation Phase Dose Level 2 (150mg Triapine) | Escalation Phase Dose Level 3 (200mg Triapine) | Expansion Phase Dose Level 1 (100mg Triapine) | Expansion Phase Dose Level 2 (150mg Triapine)
Number analyzed (Participants) | 3 | 11 | 0 | 2 | 12
percentage of participants | 33.3 | 18.2 |  | 0 | 21.4

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Will be estimated using the Kaplan-Meier curve and median estimates and confidence intervals will be calculated.
Time Frame: Time from registration to time of progressive disease as defined by Response Evaluation Criteria in Solid Tumors 1.1 criteria or death from any cause, whichever occurs first, assessed up to 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Description: Will be estimated using the Kaplan-Meier curve and median estimates and confidence intervals will be calculated.
Time Frame: The time from date of enrollment to the date of death due to any cause, assessed up to 24 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Expression of Somatostatin Receptors
Description: Will be summarized using descriptive statistics and changes from baseline versus follow-up time points will be assessed using paired test methodologies.
Time Frame: Up to 24 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Whole Exome Sequencing
Description: Will be processed using the data processing and data analysis pipelines from the Biostatistics and Bioinformatics shared resource of Markey Cancer Center to identify candidate mutated genes with adjustment for false discovery rate.
Time Frame: Up to 24 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Pharmacokinetic (PK) Studies
Description: PK parameters will be estimated from patients enrolled in the dose escalation portion of the phase 1 trial. PK parameters will be compared with historical controls, and exploratorily, we may correlate exposure to toxicity, and incorporate data into a population PK model.
Time Frame: Up to 24 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Krenning Score From the Gallium 68 Dotatate
Description: Will be summarized by calculating the proportion of patients in each Krenning score category and exploratory assessments for association with clinical response (ORR) will be performed using Fisher's exact test. Median, interquartile range will be calculated for quantitative image measurements from gallium 68 dotatate and exploratory comparison of levels with clinical response (ORR) will be performed using two sample t-test or nonparametric analogs. Correlative endpoint analyses will be based on patients who received the recommended phase 2 dose from the dose escalation portion and expansion cohort.
Time Frame: Up to 24 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Deoxyribonucleoside Concentrations
Description: Will be assessed by paired t-test or other methods. Deoxynucleoside plasma concentration as a predictor of clinical outcomes will explored by linear (progression free survival) and logistic regression (response).
Time Frame: Baseline up to 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Escalation Phase Dose Level 1 (100mg Triapine) | Escalation Phase Dose Level 2 (150mg Triapine) | Escalation Phase Dose Level 3 (200mg Triapine) | Expansion Phase Dose Level 1 (100mg Triapine) | Expansion Phase Dose Level 2 (150mg Triapine)
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/11 | 0/1 | 0/2 | 2/14
Serious Adverse Events (participants affected / at risk) | 3/3 | 8/11 | 1/1 | 2/2 | 11/14
Other Adverse Events (participants affected / at risk) | 3/3 | 11/11 | 1/1 | 2/2 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Phase Dose Level 1 (100mg Triapine) (N=3) | Escalation Phase Dose Level 2 (150mg Triapine) (N=11) | Escalation Phase Dose Level 3 (200mg Triapine) (N=1) | Expansion Phase Dose Level 1 (100mg Triapine) (N=2) | Expansion Phase Dose Level 2 (150mg Triapine) (N=14)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 4 (5)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 6 (6) | 0 (0) | 2 (2) | 8 (9)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 7 (7)
Platelet count decreased (Investigations) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 4 (4)
White blood cell decreased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 7 (7)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Phase Dose Level 1 (100mg Triapine) (N=3) | Escalation Phase Dose Level 2 (150mg Triapine) (N=11) | Escalation Phase Dose Level 3 (200mg Triapine) (N=1) | Expansion Phase Dose Level 1 (100mg Triapine) (N=2) | Expansion Phase Dose Level 2 (150mg Triapine) (N=14)
Anemia (Blood and lymphatic system disorders) | 3 (17) | 10 (51) | 0 (0) | 2 (20) | 12 (47)
Methemoglobinemia (Blood and lymphatic system disorders) | 0 (0) | 3 (16) | 0 (0) | 0 (0) | 0 (0)
Aortic Valve Disease (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (9)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (15)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (5) | 9 (30) | 1 (1) | 2 (8) | 5 (11)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 3 (5)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 1 (2) | 4 (10) | 0 (0) | 2 (13) | 2 (9)
Fatigue (General disorders) | 1 (4) | 6 (34) | 1 (1) | 2 (19) | 7 (24)
Fever (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (6) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (5) | 3 (8) | 0 (0) | 2 (5) | 2 (2)
Alkaline phosphatase increased (Investigations) | 3 (14) | 2 (8) | 0 (0) | 1 (2) | 4 (16)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (8) | 0 (0) | 1 (2) | 4 (8)
Blood bilirubin increased (Investigations) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 8 (14)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 5 (13) | 0 (0) | 2 (6) | 5 (13)
Creatinine Increased (Investigations) | 2 (2) | 4 (24) | 0 (0) | 0 (0) | 2 (4)
Investigations - Other (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Lymphocyte count decreased (Investigations) | 3 (20) | 10 (47) | 0 (0) | 2 (13) | 11 (50)
Neutrophil count decreased (Investigations) | 2 (9) | 5 (16) | 0 (0) | 1 (2) | 6 (12)
Platelet count decreased (Investigations) | 3 (14) | 6 (24) | 0 (0) | 2 (4) | 8 (33)
Weight gain (Investigations) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 1 (6)
Weight loss (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 3 (20) | 7 (28) | 0 (0) | 2 (11) | 10 (18)
Anorexia (Metabolism and nutrition disorders) | 2 (7) | 4 (9) | 0 (0) | 1 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7) | 2 (7) | 0 (0) | 1 (6) | 3 (10)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminnemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 4 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (11) | 2 (4) | 0 (0) | 1 (1) | 4 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (11)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 2 (3) | 0 (0) | 1 (3) | 3 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (10) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (6)
Paresthesia (Nervous system disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (7) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (7) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urine discolaration (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (8) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Hypertension (Vascular disorders) | 0 (0) | 3 (12) | 0 (0) | 0 (0) | 3 (11)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Eye disorders -other (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (11)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (23) | 1 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (7)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Vascular disorders - other (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT04234568/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT04234568/ICF_002.pdf